CLINICAL TRIAL: NCT05764213
Title: Improving Maternal Mental Health & Substance Use Disorder Screening and Treatment
Brief Title: Improving Maternal Mental Health & SUD Screening and Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Constance Guille, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 00123833
Record Dates: First submitted 2023-02-17; First posted 2023-03-10 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Mental Health Issue; Substance Use Disorders; Postpartum Depression; Postpartum Anxiety
MeSH Terms: conditions — Substance-Related Disorders; Depression, Postpartum | interventions — Gravidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening Brief Intervention & Referral to Treatment (SBIRT) (No Intervention): This group will receive in-person screening and referral to treatment assessment.
- Listening to Women & Pregnant & Postpartum People (LTWP) (Experimental): This group will receive text-message-based SBIRT with phone-based assessment and referral to treatment. The SBIRT is a survey with 9 questions related to depression, anxiety, substance abuse (alcohol, cigarettes, and other drugs including prescription medication), and domestic violence.
  Interventions: Behavioral: Listening to Women & Pregnant and Postpartum People

INTERVENTIONS:
Behavioral: Listening to Women & Pregnant and Postpartum People — Participants are enrolled in text message-based screenings with immediate automated feedback, paired with remote care coordination and, if appropriate, home-based telemedicine mental health and substance use disorder treatment services.
  Arms: Listening to Women & Pregnant & Postpartum People (LTWP)

SUMMARY:
The purpose of the study is to compare a text message-based mental health and substance use screening and referral to a treatment program, called Listening to Women and Pregnant and Postpartum People (LTWP), to standard of care in-person mental health and substance use screening to look at rates of treatment attendance and retention in treatment. Participation would involve completing online questionnaires. You may be eligible to participate if you are age 18-45 years, are pregnant and entering prenatal care in one of MUSC's OB clinics, and attended a prenatal appointment at an MUSC clinic.

DETAILED DESCRIPTION:
Aim 1: To determine differences in rates of treatment attendance and retention for Perinatal Mood and Anxiety Disorders (PMADs) and Perinatal Substance Use Disorders (PSUDs) between participants assigned to LTWP, compared to SBIRT.

Aim 2: To determine differences in Patient-Reported Outcomes (PROs) including depressive symptoms, quality of life, substance use, and maternal functioning and well-being measured at baseline and 2, 5, 8, and 11 months postpartum.

ELIGIBILITY:
Aim 1:

This study is a cluster RCT step wedge design so we are randomizing on the clinic level, not the individual level. The clinics are made up of 4 "wedges" (3 clinics/wedge). Pregnant women receiving prenatal care in these clinics will receive SBIRT as part of usual care. Clusters of clinics will be randomized to an LTWP start date where they will transition from SBIRT to LTWP for the purposes of screening and referral to treatment.

EHR Data Collection (PPP):

Inclusion:

1. Age 18-45
2. pregnant and entering prenatal care in one of MUSC's OB clinics
3. attended a prenatal appointment at an MUSC clinic

Exclusion:

a.) primary language is not English or Spanish

Aim 2:

Study Assessments at baseline and 2, 5, 8, and 11 months postpartum (PPP):

Inclusion:

1. Age 18-45 years
2. pregnant
3. attended an initial prenatal appointment at an MUSC OB clinic

Exclusion:

1. Unable to complete study assessments
2. primary language is not English or Spanish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10473 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Treatment Attendance | Through participants baseline prenatal care appointment and pregnancy and the postpartum year for participants, approximately 21 months
  Treatment attendance is defined as attending at least 1 or more visits with a mental health or substance use disorder treatment provider.
Change in Retention in Treatment | Through participants baseline prenatal care appointment and pregnancy and the postpartum year for participants, approximately 21 months
  Retention in treatment for PMADs: defined as 6 or more psychotherapy visits and/or 4 or more medication management visits; and PSUDs: are defined as continuous pharmacological and/or behavioral treatment > 2 months.

SECONDARY OUTCOMES:
Change in depressive symptoms | Change from baseline depression screening symptoms to follow-up depression screening symptoms during the postpartum year, approximately over 21 months.
  We will compare the mean change in the Edinburgh Postnatal Depression Scale (EPDS) among those assigned to LTWP compared to SBIRT.
  A score of 10 or more on the EPDS suggests clinically elevated depressive symptoms requiring further evaluation.
  A higher score on the EPDS is a worse outcome.
Change in Substance Use | Change from baseline substance use to follow-up substance use during the postpartum year, approximately over 21 months.
  We will compare the change in substance use frequency and amount as measured by the ASSIST among those assigned to LTWP compared to SBIRT.
  A score of 0-3 (0-4 for cannabis) has an indicated response for brief education, a score of 4-26 (5-26 for cannabis) has an indicated response for brief intervention, a score of 27+ has an indicated response for brief intervention (offer options that include treatment).
Change in Maternal Functioning and Wellbeing | Change from baseline maternal functioning to follow-up maternal functioning during the postpartum year, approximately over 21 months.
  We will compare the change in maternal functioning measured by the Barkin Index of Maternal Functioning among those assigned to LTWP compared to SBIRT.
  Each item is rated on a 7-point likert scale ranging from 0 = "strongly disagree" to 6 = "strongly agree". The total score ranges from 0 to 120. Higher levels of functioning are associated with higher total scores with 120 representing optimal functioning. Lower levels of functioning are associated with lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: Constance Guille, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States